CLINICAL TRIAL: NCT04669873
Title: Clinical Trial, Randomized, Open Label, With an Active Comparator to Assess the Efficacy and Safety of Using Accelerated Partial Irradiation Versus Standard or Hypofractionated Irradiation of the Entire Breast in Patients With Initial Breast Cancer After Conservative Surgery
Brief Title: Accelerated Partial Breast Irradiation Versus Standard or Hypofractionated Whole-Breast Irradiation, in Early Breast Cancer, After Breast-conserving Surgery
Acronym: LAPIDARY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Eduardo Barbieri, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38341220.8.0000.0072
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasm of Breast
Keywords: Breast Cancer; Radiotherapy; Hypofractionated; Breast-conserving surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: Standard (Active Comparator): Whole breast Radiotherapy, 40 Gray (40Gy) fractions
  Interventions: Radiation: Active Comparator: Standard
- Experimental 1: Hypofractionated radiotherapy (Experimental): Whole breast Radiotherapy, 26 Gray (26Gy) in 5 fractions
  Interventions: Radiation: Experimental 1: Hypofractionated radiotherapy
- Experimental 2: Accelerated Partial Breast Irradiation (Experimental): Partial Breast Irradiation 26 Gray (26Gy) to the tumor bed in 5 fractions.
  Interventions: Radiation: Experimental 2: Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: Active Comparator: Standard — Radiation: Whole Breast Irradiation + Boost Whole breast, either 40Gy, in 15 fractions, in 3 weeks
  Arms: Active Comparator: Standard
Radiation: Experimental 1: Hypofractionated radiotherapy — Radiation: Hypofractionated irradiation Whole Breast Irradiation 26Gy in 5 fractions in one week
  Arms: Experimental 1: Hypofractionated radiotherapy
Radiation: Experimental 2: Accelerated Partial Breast Irradiation — Radiation: Accelerated partial breast irradiation Tumor bed 26Gy in 5 fractions, in 5 days.
  Arms: Experimental 2: Accelerated Partial Breast Irradiation

SUMMARY:
Radiotherapy has been confirmed as an important treatment breast-conserving surgery reducing the risk of any recurrence of breast cancer and breast cancer-related mortality in patients with early breast cancer.

There are no comparative data on the ideal radiotherapy treatment regimen for patients with early stage breast cancer who underwent conservative surgery in the Brazilian population.

DETAILED DESCRIPTION:
The investigators propose a prospective, randomized, pilot study, with active control, to evaluate the viability and safety of accelerated partial breast irradiation, in 5 fractions, comparing with the radiotherapy regimens of the whole breast in 15 and 5 fractions, in patients with breast cancer, in initial stage, who underwent conservative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Information to the patient and signed informed consent;
* Women aged ≥50 years
* Breast conserving surgery
* Pathologic tumor size < 3 cm (maximum microscopic diameter of the invasive component)
* Invasive adenocarcinoma (except classic invasive lobular carcinoma)
* Unifocal disease
* Histopathologic grades I or II
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Lymphovascular invasion absent
* Negative axillary lymph nodes
* Minimum microscopic margins of non-cancerous tissue of 2mm (excluding deep margin when in deep fascia)
* No prior breast or mediastinal radiotherapy
* No hematogenous metastases

Exclusion Criteria:

* Previous malignancy (except non-melanomatous skin cancer)
* Mastectomy
* Classical-Type Invasive Lobular Carcinoma
* Neoadjuvant chemotherapy
* Human Epidermal growth factor Receptor-type 2 positive (HER2+)
* Triple-negative breast cancers
* Intravascular lymphoma present
* Contraindications to radiotherapy.
* No geographical, social or psychologic reasons that would prevent study follow

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of local recurrence | 5 years
  To estimate and compare the rate of local recurrence between the experimental and control arms.

SECONDARY OUTCOMES:
Time to occurrence of distant metastases | 5 years
  Distant tumor time is defined as number of days from randomization until occurrence of distant metastases, death without prior distant progression, or end of follow-up.
Disease-free survival | 5 years
  Disease-free survival, defined as number of days from randomization until the first occurrence of local recurrence, distant metastases, tumor-related death, death without prior progression, or end of follow-up.
Overall survival | 5 years
  Overall survival time, defined as number of days from randomization until death or end of follow-up.
Medico-economic study | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate and compared the cost between Accelerated Partial Breast Irradiation with Standard and Hypofractionated irradiation
Health-related Quality of Life | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate the patients quality of life with the help of the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). This questionnaire was designed to be cancer specific, multidimensional in structure, suitable for self-administration (brief and easy to complete), and applicable in a wide range of cultural contexts. The scores in each dimension are uniformly transformed to dimensions ranging from 0 to 100, with 0 denoting the negative (low functioning, high symptom burden) and 100 the positive end (high functioning, low symptom burden) of the continuum.
Evaluation of quality of life change by European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate the patient quality of life with the help of the European Organization for Research and Treatment of Cancer Breast-Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23). The 23-item EORTC QLQ BR23 contains two breast cancer specific functional scales (body image and sexuality) and three symptom scales evaluating arm symptoms, breast symptoms, and systemic therapy symptoms. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Fatigue Questionnaire (Functional Assessment of Cancer Therapy-Fatigue - FACT-F) | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate the patient quality of life with the help of the Functional Assessment of Cancer Therapy-Fatigue (FACT-F). Scores are interpreted according to the guidelines of the Scoring Manual. The higher the number of points, the better the quality of life. To obtain the score, the negative questions are reverted; then the answers of the domains are added up, and a proportional average is carried out in case of non answered items.
Measurement Satisfaction of Body Image of the participants | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate the patient quality of life and patient satisfaction with the help of the Body Image Scale (BIS). Scores are interpreted according to the guidelines of the Scoring Manual. The Body Image Scale (BIS) is a self-assessment scale designed to assess cancer patients' perceptions of their appearance and identify any changes to those perceptions resulting from a disease or a treatment. The total score ranges from 0 to 30. A higher score means a higher level of body image disturbance.
Changes in anxiety and depression | Baseline and 3 months, 6 months, 12 months, 2 years, 5 years after treatment end
  To evaluate the patient quality of life and patient satisfaction with the help of the Hospital Anxiety and Depression Scale (HADS). Scores for each sub scale (depression and anxiety) are summed-up and range from 0 to 21. Values from 0-7 indicate normal levels, 8-10 are border values and values from 11-21 are considered to be pathological.
Early and late adverse effects in normal tissues | 5 years
  To evaluate the results reported by patient and evaluated by doctors, as well as, photographic assessments.
Late adverse effects | 5 years
  To evaluate if the patient had symptoms of swelling or edema in the arm, breast shrinkage, hardness, pigmentation, necrosis, pain and tenderness in the breast.
Acute toxicity rate | 5 years
  To evaluate acute toxicity rate. The maximum grade for acute toxicity will be recorded for each patient at each treatment evaluation using Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Locations (1):
- IBCC Oncologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The findings will be shared and discussed with all investigators in the study. A study manuscript, having received contributions from all authors, will be submitted for publication in scientific circles.

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Darby S, McGale P, Correa C, Taylor C, Arriagada R, Clarke M, Cutter D, Davies C, Ewertz M, Godwin J, Gray R, Pierce L, Whelan T, Wang Y, Peto R. Effect of radiotherapy after breast-conserving surgery on 10-year recurrence and 15-year breast cancer death: meta-analysis of individual patient data for 10,801 women in 17 randomised trials. Lancet. 2011 Nov 12;378(9804):1707-16. doi: 10.1016/S0140-6736(11)61629-2. Epub 2011 Oct 19. PMID 22019144
- [Background] Strnad V, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Hindemith M, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). 5-year results of accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy versus whole-breast irradiation with boost after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: a randomised, phase 3, non-inferiority trial. Lancet. 2016 Jan 16;387(10015):229-38. doi: 10.1016/S0140-6736(15)00471-7. Epub 2015 Oct 19. PMID 26494415
- [Background] Polgar C, Fodor J, Major T, Sulyok Z, Kasler M. Breast-conserving therapy with partial or whole breast irradiation: ten-year results of the Budapest randomized trial. Radiother Oncol. 2013 Aug;108(2):197-202. doi: 10.1016/j.radonc.2013.05.008. Epub 2013 Jun 3. PMID 23742961
- [Background] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717
- [Background] Correa C, Harris EE, Leonardi MC, Smith BD, Taghian AG, Thompson AM, White J, Harris JR. Accelerated Partial Breast Irradiation: Executive summary for the update of an ASTRO Evidence-Based Consensus Statement. Pract Radiat Oncol. 2017 Mar-Apr;7(2):73-79. doi: 10.1016/j.prro.2016.09.007. Epub 2016 Sep 17. PMID 27866865
- [Background] Livi L, Meattini I, Marrazzo L, Simontacchi G, Pallotta S, Saieva C, Paiar F, Scotti V, De Luca Cardillo C, Bastiani P, Orzalesi L, Casella D, Sanchez L, Nori J, Fambrini M, Bianchi S. Accelerated partial breast irradiation using intensity-modulated radiotherapy versus whole breast irradiation: 5-year survival analysis of a phase 3 randomised controlled trial. Eur J Cancer. 2015 Mar;51(4):451-463. doi: 10.1016/j.ejca.2014.12.013. Epub 2015 Jan 17. PMID 25605582
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Background] Brunt AM, Haviland JS, Sydenham M, Agrawal RK, Algurafi H, Alhasso A, Barrett-Lee P, Bliss P, Bloomfield D, Bowen J, Donovan E, Goodman A, Harnett A, Hogg M, Kumar S, Passant H, Quigley M, Sherwin L, Stewart A, Syndikus I, Tremlett J, Tsang Y, Venables K, Wheatley D, Bliss JM, Yarnold JR. Ten-Year Results of FAST: A Randomized Controlled Trial of 5-Fraction Whole-Breast Radiotherapy for Early Breast Cancer. J Clin Oncol. 2020 Oct 1;38(28):3261-3272. doi: 10.1200/JCO.19.02750. Epub 2020 Jul 14. PMID 32663119
- [Background] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Background] Imielinski K. [Sexuality and personality]. Ginekol Pol. 1981 Mar;52(3):293-7. No abstract available. Polish. PMID 7262592